CLINICAL TRIAL: NCT02410616
Title: European Comparative Effectiveness Research on Internet-based Depression Treatment - Swiss Trial
Brief Title: E-Compared-CH: Comparative Effectiveness Research on Internet-based Depression Treatment - Swiss Trial
Acronym: E-COMPARED_CH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001/15
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Depressive Disorder, Major
Keywords: Psychotherapy; Comparative Effectiveness Research; Randomized Controlled Trial; Secondary Care
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blended CBT (Experimental): Internet based blended CBT depression treatment combines individual face-to-face cognitive behavioural therapy (CBT) with CBT delivered through an Internet based treatment platform with mobile phone components. The core components of the CBT treatment are: (1) psychoeducation, (2) behavioural activation, (3) cognitive restructuring, and (4) relapse prevention.
  Interventions: Behavioral: Blended CBT
- Treatment as usual (Active Comparator): Treatment as usual (TAU) is defined as the routine care that subjects receive when they are diagnosed with depression in the secondary care system. The investigators will not interfere with treatment as usual but they will monitor carefully which health care services are utilized by usual care patients using patient records and through self-report.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Blended CBT — Internet based blended CBT depression treatment combines individual face-to-face cognitive behavioural therapy (CBT) with CBT delivered through an Internet based treatment platform with mobile phone components. The core components of the CBT treatment are: (1) psychoeducation, (2) behavioural activation, (3) cognitive restructuring, and (4) relapse prevention.
  Arms: Blended CBT
Behavioral: Treatment as usual — Treatment as usual (TAU) is defined as the routine care that subjects receive when they are diagnosed with depression in the secondary care system. The investigators will not interfere with treatment as usual but they will monitor carefully which health care services are utilized by usual care patients using patient records and through self-report.
  Arms: Treatment as usual

SUMMARY:
To compare the clinical and cost-effectiveness of blended Cognitive Behavioural Therapy (CBT) for adults with major depressive disorder (MDD) with treatment as usual (TAU) in Swiss patients in secondary care

DETAILED DESCRIPTION:
Background

Depression is a common mental disorder with a negative impact on mental well-being, quality of life, and social and work-related functioning both in the short and longer term. Additionally, depression is associated with increased morbidity, mortality, health care utilization and health care costs. On a population level, depression is one of the most costly diseases. The economic costs of depression were estimated at €136.3 billion (EU25) in 2010 in the EU and are still rising. European health care systems face the challenge of improving access to cost-effective treatments while simultaneously working to sustain budgetary stability in times of economic austerity.

Internet-based depression treatment appears a very promising alternative to current routine depression treatment strategies. Meta-analyses have demonstrated the clinical effectiveness and potential cost-effectiveness of Internet-based treatment for depression in controlled research setting. Internet-based treatment thus has the potential to keep depression treatment affordable, as it enables mental health care providers to reach out to large populations needing depression treatment at a better cost-effectiveness than those of standard treatment as usual (TAU), but with similar levels of clinical efficacy and quality of care. The trials will be conducted in 8 European countries.

Objective

To compare the clinical and cost-effectiveness of blended CBT and TAU in secondary care

Methods

In Switzerland, a randomized-controlled trial will be carried out in secondary care, comparing the clinical and cost-effectiveness of CBT and TAU for adults with major depressive disorder (MDD). Respondents will be followed until 12 months after baseline (measures will be taken at BL, 12 weeks, 18 weeks, 6 months and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Meet DSM-IV diagnostic criteria for MDD confirmed by MINI International Neuropsychiatric Interview version 5.0
* Informed Consent
* Having access to a PC and Internet connection
* Having a Smartphone that is compatible with the mobile component of the intervention
* Understanding of the German language spoken and written

Exclusion Criteria

* Current high risk for suicide according to the MINI Interview section C
* Serious psychiatric co-morbidity: substance dependence, bipolar affective disorder, psychotic illness, obsessive compulsive disorder, as established at the MINI interview
* Currently receiving psychological treatment for depression
* Being unable to comprehend the spoken and written language (German)
* Not having access to a PC and fast Internet connection (i.e. broadband or comparable).
* Not having a Smartphone that is compatible with the mobile component of the intervention that is offered or not willing to carry a Smartphone during the duration of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | 18 weeks

SECONDARY OUTCOMES:
Assessment of Quality of Life (AQoL-6D) | Baseline, 12 weeks, 18 weeks, 6 months, and 12 months
Quick Inventory of Depressive Symptomatology Self-Report (QIDS-16-SR) | Baseline, 12 weeks, 18 weeks, 6 months, and 12 months
MINI International Neuropsychiatric Interview (M.I.N.I; Ackenheil et al., 1999) | Baseline, 18 weeks, and 12 months
EuroQoL (EQ-5D-5L; Herdman et al., 2011) | Baseline, 12 weeks, 18 weeks, 6 months, and 12 months
Questionnaires on Costs Associated with Psychiatric Illness (TiC-P; Hakkaart-van Rooijen, van Straten, Donker, Tiemens, 2002) | Baseline, 12 weeks, 18 weeks, 6 months, and 12 months
Client Satisfaction Questionnaire (CSQ-8; Nguyen, Attkinson, & Stegner, 1983) | 12 weeks, and 18 weeks
System Usability Scale (SUS; Brooke, 1996) | 12 weeks, and 18 weeks
Patient Health Questionnaire-9 (PHQ-9) | Baseline, 12 weeks, 6 months, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Berger, PhD, Principal Investigator — University of Bern
Locations (2):
- Switzerland (2):
  - Sanatorium Kilchberg, Kilchberg, Canton of Zurich
  - Department of Clinical Psychology and Psychotherapy, Bern

REFERENCES:
- [Derived] Doukani A, Quartagno M, Sera F, Free C, Kakuma R, Riper H, Kleiboer A, Cerga-Pashoja A, van Schaik A, Botella C, Berger T, Chevreul K, Matynia M, Krieger T, Hazo JB, Draisma S, Titzler I, Topooco N, Mathiasen K, Vernmark K, Urech A, Maj A, Andersson G, Berking M, Banos RM, Araya R. Comparison of the Working Alliance in Blended Cognitive Behavioral Therapy and Treatment as Usual for Depression in Europe: Secondary Data Analysis of the E-COMPARED Randomized Controlled Trial. J Med Internet Res. 2024 May 31;26:e47515. doi: 10.2196/47515. PMID 38819882
- [Derived] van Genugten CR, Schuurmans J, Hoogendoorn AW, Araya R, Andersson G, Banos R, Botella C, Cerga Pashoja A, Cieslak R, Ebert DD, Garcia-Palacios A, Hazo JB, Herrero R, Holtzmann J, Kemmeren L, Kleiboer A, Krieger T, Smoktunowicz E, Titzler I, Topooco N, Urech A, Smit JH, Riper H. Examining the Theoretical Framework of Behavioral Activation for Major Depressive Disorder: Smartphone-Based Ecological Momentary Assessment Study. JMIR Ment Health. 2021 Dec 6;8(12):e32007. doi: 10.2196/32007. PMID 34874888
- [Derived] Kleiboer A, Smit J, Bosmans J, Ruwaard J, Andersson G, Topooco N, Berger T, Krieger T, Botella C, Banos R, Chevreul K, Araya R, Cerga-Pashoja A, Cieslak R, Rogala A, Vis C, Draisma S, van Schaik A, Kemmeren L, Ebert D, Berking M, Funk B, Cuijpers P, Riper H. European COMPARative Effectiveness research on blended Depression treatment versus treatment-as-usual (E-COMPARED): study protocol for a randomized controlled, non-inferiority trial in eight European countries. Trials. 2016 Aug 3;17(1):387. doi: 10.1186/s13063-016-1511-1. PMID 27488181